CLINICAL TRIAL: NCT03169868
Title: A Pilot Prospective, Randomized Controlled Trial Assessing Enhanced Medication Reconciliation With a Clinical Decision Support Tool in Patients With Serious Mental Illness.
Brief Title: Enhanced Medication Reconciliation For Serious Mental Illness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment rate insufficient to fully enroll study within the planned timeline.
Sponsor: Precera Bioscience, Inc. (Industry)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SAN_UPMC_Psych_001
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Mental Disorders
Keywords: clinical decision support; drug levels in blood; therapeutic drug monitoring; medication adherence; medication therapy management
MeSH Terms: conditions — Mental Disorders; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Medication reconciliation (Experimental): Medication reconciliation with pharmacist using electronic health records, pharmacy dispensing data and Sano Patient Medication Profile(TM)
  Interventions: Diagnostic Test: Sano Patient Medication Profile
- Standard Medication reconciliation (No Intervention): Medication reconciliation with pharmacist using electronic health records and pharmacy dispensing data only

INTERVENTIONS:
Diagnostic Test: Sano Patient Medication Profile — The Sano Patient Medication Profile (PMP) is a graphical report comparing prescribed medications to LC/MS/MS-detected drugs from patient blood samples
  Arms: Enhanced Medication reconciliation

SUMMARY:
The purpose of this study is to evaluate the clinical utility of a decision support tool, the Patient Medication Profile(TM), developed by Sano Informed Prescribing on medication reconciliation and identification of drug-related problems in patients with serious mental illness.

DETAILED DESCRIPTION:
Lack of adherence to medications is an identifiable and growing problem in the United States and can result in disease progression, disease complications, treatment failure, a lower quality of life, and increased morbidity and mortality. Medication-related problems and medication nonadherence have been estimated to cost $177 billion annually in total direct and indirect U.S. health care costs. Moreover, medication adherence rates are poor for individuals diagnosed with chronic conditions such as diabetes, depression, and schizophrenia, which require long-term therapy. Recent publications have estimated that nearly 50% of patients in the U.S. being treated for chronic conditions are non-adherent to their medication regimens. Although increased medication adherence may lead to increased spending on drug therapy, it is associated with greatly reduced total health care costs and usage, and better patient outcomes.

Persons diagnosed with serious mental illness (SMI) such as schizophrenia and bipolar disorder are at higher risk than the general population for medication nonadherence, cardiovascular mortality, and medical co-morbidities such as diabetes, hypertension, dyslipidemia, obesity, nicotine dependence, and coronary heart disease. Poor adherence to complex medication regimens, decreased access to care, and uncoordinated care between psychiatry and medical care teams, have been identified as key contributors to the disparities experienced by this patient population.

The United States healthcare system is complex and healthcare is fragmented, particularly for those with serious mental illness who are often prescribed multiple medications from numerous providers. One unifying piece of information that is of critical importance for optimizing patient care is the patient medication list. Unfortunately, appropriate medication reconciliation to obtain the correct medication list and information about medication adherence is a complex and imperfect process. Using patient pharmacy records, electronic health record (EHR), and patient interviews, discrepancies have been found with over one third of patients upon hospital admission. Therefore, it can be expected that most polypharmacy patients (defined as taking five or more medications) have errors in their medical record.

National and world health associations have identified several opportunities for health professionals to provide services that aim to increase medication adherence and decrease medication related problems. Several of the recommendations emphasize the use of coordinated multidisciplinary efforts to provide patients with the most access to care and the highest quality education about their medications. Pharmacists are among the most accessible health care professionals and have specialized training to identify, prevent, and resolve drug-related problems (DRPs). As medication experts, pharmacists are important members of the multidisciplinary team and are uniquely positioned to impact medication-related health outcomes through accurate medication reconciliation, comprehensive mediation reviews (CMR), and interventions to improve medication safety and adherence.

An objective measure of what medications patients are actually taking would enable healthcare teams to better identify and tailor interventions to each specific patient situation. Using a novel therapeutic drug monitoring assay and empirical clinical decision support tool, Sano has shown that errors in patient medication lists are prevalent and poorly reflect patient adherence to the intended medication regimen and actual medication exposure. For example, in a cohort of psychiatry patients, only 37% were fully adherent to all medications in their treatment regimen and roughly one in five medications detected was not in the medical record. We anticipate that when medication reconciliation is performed by a pharmacist using Sano's clinical decision support tool, medication adherence will improve and more drug therapy problems will be identified and resolved. As a result, we expect to see an improvement in patient outcomes and a reduction in healthcare spending (i.e. post-hospitalization unplanned healthcare utilization).

ELIGIBILITY:
Inclusion Criteria:

* Current insurer is UPMC Health Plan
* Currently active in CRS clinic
* Prescribed four or more medications as indicated by pre-study Health Plan Medication List
* Able to provide informed consent for present study

Exclusion Criteria:

* Not competent to give informed consent in the opinion of the investigator
* Having had a previous medication reconciliation by the clinical pharmacist

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Medical record accuracy | 3 months
  The "Final Medication List" (medications in EHR at final visit) will be compared to the detected medications as summarized in the Patient Medication Profile at final visit (approx 3 months). For each patient, the proportion of detected medications that are not in the medication list will be calculated, excluding OTC medications from the analysis. Medical record accuracy in the intervention and control groups will be compared.

SECONDARY OUTCOMES:
Automated vs. manual pharmacist-led medication reconciliation | 0 months
  Compare automated Sano Patient Medication Profile medication list to the manual pharmacist-led reconciliation which includes review of medication lists from available EHRs, pharmacy dispensing data and patient interview. For each patient in the control group, calculate the number of drug additions and/or subtractions to arrive at the "Informed Medication List" (review of EHR and pharmacy dispensing during patient interview with/without the Sano test) from the "Reconciled Medication List" (EHR, pharmacy dispensing) vs. the number of additions / subtractions to arrive at the Informed Medication List from the Patient Medication Profile.
Drug Related Problem Identification and resolution | 3 months
  Documented drug related problems identified by the pharmacist will be compared between the intervention and control groups at baseline and final visit. The number of changes in medications to resolve drug related problems, such as medication additions, terminations, dosage or frequency changes will be compared between the intervention and control groups
Adherence to prescribed medications | 3 months
  For each patient, the proportion of medications that are in the "Optimized Medication List" (medications that patient should be taking after pharmacist medication reconciliation and interview) and detected as summarized in the Patient Medication Profile will be calculated. Medications with half-life < three hours will be excluded, as will be medications prescribed "as needed" (PRN).

CONTACTS AND LOCATIONS:
Locations (1):
- Western Psychiatric Institute and Clinic of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided